CLINICAL TRIAL: NCT01039168
Title: Reduction of Person-job Mismatch to Increase Work Capacity, by Education of, and Dialogue Between Involved Parties - Evaluation of an Intervention Program
Brief Title: Return to Work After a Workplace-oriented Intervention for Patients on Sick Leave Due to Burnout
Acronym: ADA model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other); Lund University (Other); County Councils of Southern Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FAS 2003-0765
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Professional Burnout
Keywords: Burnout; Sick leave; Intervention study; Prospective study; Work
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Workplace dialogue (Active Comparator): Clinical examination and dialogue with supervisor to find solutions to reduce job-person mismatch and facilitate return to work
  Interventions: Behavioral: Workplace dialogue
- Care as usual (Sham Comparator): No intervention besides of the care as usual being available for the patient
  Interventions: Other: Care as usual

INTERVENTIONS:
Behavioral: Workplace dialogue
  Arms: Workplace dialogue
Other: Care as usual
  Arms: Care as usual

SUMMARY:
The study aims to evaluate the effect on return to work of a workplace intervention with patients being treated for burnout. The intervention intends to reduce job-person mismatch through patient-supervisor communication.The hypothesis is that the intervention group will show a more favourable outcome than a control group with respect to return to work.

DETAILED DESCRIPTION:
Participants are consecutively recruited in co-operation with regional social insurance offices (RSIOs) in the two southern counties of Sweden. Persons accepting participation are clinically examined and interviewed of the course of events leading up to the burnout and the patient's expectations of changes necessary to facilitate return to work are recorded. The patient´s supervisor is then interviewed at the workplace, responding to the same questions on perceived main causes of the subordinate's sick leave and changes necessary to facilitate return to work. Finally, the core intervention takes place, namely a dialogue being initiated between the patient and the supervisor to find solutions to facilitate return to work. Out of those who do not want to participate, without giving any specific reason for that, a control group is matched by length and degree of sick leave at the time of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* employment
* sick leave at lest half time 2-6 months due to work related burnout
* previously healthy

Exclusion Criteria:

* other somatic or psychiatric disease explaining the symptoms

Max Age: 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2003-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Return to work from sick leave | Up to 1,5 years post intervention completion

SECONDARY OUTCOMES:
Self-rated health measures (only in the intervention group) | Up to 1,5 years post intervention completion

CONTACTS AND LOCATIONS:
Overall Officials: Björn Karlson, PhD, Principal Investigator — Occupational and Environmental Medicine, Lund University Hospital and Lund University
Locations (1):
- Occupational and Environmental Medicine, Lund University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Karlson B, Jonsson P, Palsson B, Abjornsson G, Malmberg B, Larsson B, Osterberg K. Return to work after a workplace-oriented intervention for patients on sick-leave for burnout--a prospective controlled study. BMC Public Health. 2010 Jun 2;10:301. doi: 10.1186/1471-2458-10-301. PMID 20515510